CLINICAL TRIAL: NCT02863861
Title: Comparative Study Between Propofol-Ketamine Combination and Dexmedetomidine-Ketamine Combination for Sedation in Upper Gastrointestinal Endoscopy in Paediatric Patients.
Brief Title: Sedation for Upper Gastrointestinal Endoscopy in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Akram Mohamed Mohamed Amer, Lecturer in Department of Anesthesiology, Intensive Care, and Pain Management, Faculty of Medicine, Ain-Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: FMASU R 12/2016
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Upper Gastrointestinal Endoscopy
Keywords: Sedation; Pediatric Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Group PK (Experimental): Propofol-Ketamine group: patients in this group will receive IV ketamine at a dose of 1mg.kg-1 in addition to IV propofol 1mg.kg-1 for induction with added doses of propofol 1mg.kg-1 when needed.
  Interventions: Drug: propofol-ketamine
- Group DK (Experimental): Dexmedetomidine-Ketamine group: patients in this group will receive IV ketamine at a dose of 1mg.kg-1 in addition to IV dexmedetomidine 0.5 mcg.kg-1 for induction with additional doses of dexmedetomidine 0.5mcg.kg-1 when required
  Interventions: Drug: Dexmedetomidine-ketamine

INTERVENTIONS:
Drug: Dexmedetomidine-ketamine
  Arms: Group DK
Drug: propofol-ketamine
  Arms: Group PK

SUMMARY:
The purpose of this study is to compere between Propofol-Ketamine combination and Dexmedetomidine-Ketamine combination for sedation in upper gastrointestinal endoscopy in paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists ASA I-II patients aging 2-7 years.

Exclusion Criteria:

known allergy to any of the study drugs, significant cardiovascular disease vomiting.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
length of stay in PACU | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university- faculty of medicine- department of anesthesia, intensive care and pain management, Cairo, Egypt

REFERENCES:
- [Derived] Amer AM, Youssef AM, El-Ozairy HS, El-Hennawy AM. [Propofol-ketamine versus dexmedetomidine-ketamine for sedation during upper gastrointestinal endoscopy in pediatric patients: a randomized clinical trial]. Braz J Anesthesiol. 2020 Nov-Dec;70(6):620-626. doi: 10.1016/j.bjan.2020.08.005. Epub 2020 Dec 5. PMID 33293038